CLINICAL TRIAL: NCT06307652
Title: A Phase III, Randomised, Double-blind Study to Evaluate the Effect of Balcinrenone/Dapagliflozin, Compared With Dapagliflozin, on the Risk of Heart Failure Events and Cardiovascular Death in Patients With Heart Failure and Impaired Kidney Function
Brief Title: Study to Evaluate the Effect of Balcinrenone/Dapagliflozin in Patients With Heart Failure and Impaired Kidney Function
Acronym: BalanceD-HF
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6402C00012; 2023-508162-15-00 (Registry Identifier: EU CT number)
Record Dates: First submitted 2024-02-06; First posted 2024-03-13 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure and Impaired Kidney Function
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Intervention Model Description: international, multi-centre, randomised, double-blind, parallel-group, double-dummy, active-controlled, event-driven
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- balcinrenone/dapagliflozin 15 mg/10 mg (Experimental): Patients will be randomized 1:1:1 to either combination of balcinrenone/dapagliflozin and matching placebo for dapagliflozin or dapagliflozin and matching placebo for balcinrenone/dapagliflozin
  Interventions: Drug: balcinrenone/dapagliflozin 15 mg/10 mg and matching placebo for dapagliflozin 10 mg
- balcinrenone/dapagliflozin 40 mg/10 mg (Experimental): Patients will be randomized 1:1:1 to either combination of balcinrenone/dapagliflozin and matching placebo for dapagliflozin or dapagliflozin and matching placebo for balcinrenone/dapagliflozin
  Interventions: Drug: balcinrenone/dapagliflozin 40 mg/10 mg and matching placebo for dapagliflozin 10 mg
- dapagliflozin 10 mg (Active Comparator): Patients will be randomized 1:1:1 to either combination of balcinrenone/dapagliflozin and matching placebo for dapagliflozin or dapagliflozin and matching placebo for balcinrenone/dapagliflozin
  Interventions: Drug: dapagliflozin 10 mg and matching placebo for balcinrenone/dapagliflozin

INTERVENTIONS:
Drug: balcinrenone/dapagliflozin 15 mg/10 mg and matching placebo for dapagliflozin 10 mg — 1 capsule of balcinrenone/dapagliflozin 15 mg/10 mg and 1 tablet of matching placebo for dapagliflozin 10 mg once daily, oral use
  Arms: balcinrenone/dapagliflozin 15 mg/10 mg
Drug: balcinrenone/dapagliflozin 40 mg/10 mg and matching placebo for dapagliflozin 10 mg — 1 capsule of balcinrenone/dapagliflozin 40 mg/10 mg and 1 tablet of matching placebo for dapagliflozin 10 mg once daily, oral use
  Arms: balcinrenone/dapagliflozin 40 mg/10 mg
Drug: dapagliflozin 10 mg and matching placebo for balcinrenone/dapagliflozin — 1 tablet of dapagliflozin 10 mg and 1 capsule of matching placebo for balcinrenone/dapagliflozin once daily, oral use
  Arms: dapagliflozin 10 mg

SUMMARY:
This is a Phase III, international, multi-centre, randomised, double-blind, parallel-group, double-dummy, active-controlled, event-driven study in patients with chronic HF and impaired kidney function who had a recent HF event. The aim is to evaluate the effect of balcinrenone/dapagliflozin vs dapagliflozin, given once daily on top of other classes of SoC, on CV death and HF events.

DETAILED DESCRIPTION:
The purpose of this study is to investigate the effect of balcinrenone/dapagliflozin compared with dapagliflozin, on the risk of CV death, HF event with and without hospitalisation, in patients with chronic HF, impaired kidney function, and who have had a recent HF event.

Eligible patients will randomly be assigned with a 1:1:1 ratio to receive once daily administration of one capsule and one tablet of one of the following treatments:

1. Balcinrenone/dapagliflozin 15 mg/10 mg capsule and matching placebo for dapagliflozin 10 mg tablet
2. Balcinrenone/dapagliflozin 40 mg/10 mg capsule and matching placebo for dapagliflozin 10 mg tablet
3. Dapagliflozin 10 mg tablet and matching placebo for balcinrenone/dapagliflozin capsule

The study is event driven, and the average study duration for a participant is estimated to be 22 months including screening period, 20 months blinded treatment period and a one-month follow-up period on open-label dapagliflozin.

The study will be conducted at approximately 700 sites in approximately 40 countries globally.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Documented diagnosis of symptomatic HF (NYHA functional class II-IV)
* Having had a recent HF event within 6 months (hospitalization or urgent visit)
* Have a LVEF value from an assessment within the last 12 months
* Managed with SoC therapy for HF and renal impairment according to local guidelines
* NT-proBNP must be >300 pg/mL (>600 pg/mL if concomitant atrial fibrillation or atrial flutter)
* Not taking an MRA
* An eGFR ≥ 20 to < 60 mL/min/1.73 m2
* Serum/plasma potassium ≤ 5.0 mmol/L

Exclusion Criteria:

* Acute coronary syndrome (unstable angina or myocardial infarction), stroke or transient ischaemic attack within the previous 3 months prior to enrolment or during the screening period
* Major cardiac surgery, coronary revascularisation or valvular repair or replacement, or implantation of a Cardiac resynchronisation therapy device within 3 months prior to enrolment or during the screening period, or planned to undergo any of these operations
* History of hypertrophic obstructive cardiomyopathy
* Complex congenital heart disease or severe uncorrected primary valvular disease
* Symptomatic bradycardia or second- or third-degree heart block without a pacemaker
* Systolic BP < 90 mmHg, or symptomatic hypotension within the past 24 hours
* Primary pulmonary hypertension, chronic pulmonary embolism, severe pulmonary disease including COPD or exacerbation of COPD requiring invasive mechanical ventilation assistance within 12 months prior to enrolment
* Type 1 diabetes mellitus
* Kidney replacement therapy in the past 4 weeks, currently requiring kidney replacement or imminent plan to start kidney replacement therapy
* Acute or chronic liver disease with severe impairment of liver function, eg, ascites, oesophageal varices, coagulopathy, and encephalopathy
* Suspected or confirmed COVID-19 infection within the last 4 weeks or hospitalisation for COVID-19 within the last 12 weeks
* Treatment with strong or moderate CYP3A4 inhibitor or inducer

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4800 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2027-06-11 (Estimated); Study Completion 2027-06-11 (Estimated)

PRIMARY OUTCOMES:
Time to first occurrence of any of the components of the composite of: •CV death •HF hospitalisation •HF event without hospitalisation | Approximately 38 months
  To determine whether balcinrenone/dapagliflozin is superior to dapagliflozin in reducing the risk of CV death and HF events with and without hospitalisation

SECONDARY OUTCOMES:
Total occurrences (first and recurrent) of the components of the composite of: •CV death •HF hospitalisation •HF event without hospitalisation | Approximately 38 months
  To determine whether balcinrenone/dapagliflozin is superior to dapagliflozin in reducing the rate of total occurrences of CV death, and HF events with and without hospitalisation
Total occurrences (first and recurrent) of HF hospitalisations | Approximately 38 months
  To determine whether balcinrenone/dapagliflozin is superior to dapagliflozin in reducing the rate of total HF hospitalisations
Time to CV death | Approximately 38 months
  To determine whether balcinrenone/dapagliflozin is superior to dapagliflozin in reducing the risk of CV death
The hierarchical composite endpoint of death from any cause, total HF events, and change from baseline in KCCQ total symptom score to 24-week post-randomisation | Approximately 24 weeks
  To determine whether balcinrenone/dapagliflozin is superior to dapagliflozin in reducing the risk of death from any cause, HF events, and improving patient reported symptoms of HF
Time to death from any cause | Approximately 38 months
  To determine whether balcinrenone/dapagliflozin is superior to dapagliflozin in reducing the risk of death from any cause

CONTACTS AND LOCATIONS:
Locations (644):
- United States (145):
  - Research Site, Alexander City, Alabama
  - Research Site, Birmingham, Alabama
  - Research Site, Fairhope, Alabama
  - Research Site, Huntsville, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, Beverly Hills, California
  - Research Site, Covina, California
  - Research Site, Encinitas, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Redding, California
  - Research Site, San Diego, California
  - Research Site, San Francisco, California
  - Research Site, Santa Ana, California
  - Research Site, Thousand Oaks, California
  - Research Site, Vista, California
  - Research Site, West Hills, California
  - Research Site, Aurora, Colorado
  - Research Site, Wheat Ridge, Colorado
  - Research Site, Altamonte Springs, Florida
  - Research Site, Boca Raton, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Palm Beach Gardens, Florida
  - Research Site, Pensacola, Florida
  - Research Site, Port Charlotte, Florida
  - Research Site, Safety Harbor, Florida
  - Research Site, Saint Augustine, Florida
  - Research Site, St. Petersburg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Peachtree City, Georgia
  - Research Site, Thomasville, Georgia
  - Research Site, Tucker, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Glenview, Illinois
  - Research Site, Hazel Crest, Illinois
  - Research Site, North Chicago, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Winfield, Illinois
  - Research Site, Elkhart, Indiana
  - Research Site, Evansville, Indiana
  - Research Site, Hammond, Indiana
  - Research Site, Indianapolis, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Munster, Indiana
  - Research Site, Richmond, Indiana
  - Research Site, Waterloo, Iowa
  - Research Site, Wichita, Kansas
  - Research Site, Louisville, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, West Monroe, Louisiana
  - Research Site, Augusta, Maine
  - Research Site, Rockville, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Fall River, Massachusetts
  - Research Site, Worcester, Massachusetts
  - Research Site, Ann Arbor, Michigan
  - Research Site, Bloomfield Hills, Michigan
  - Research Site, Dearborn, Michigan
  - Research Site, Farmington Hills, Michigan
  - Research Site, Flint, Michigan
  - Research Site, Troy, Michigan
  - Research Site, Ypsilanti, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, Saint Paul, Minnesota
  - Research Site, Jackson, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, Lincoln, Nebraska
  - Research Site, Las Vegas, Nevada
  - Research Site, North Las Vegas, Nevada
  - Research Site, Bridgewater, New Jersey
  - Research Site, Jersey City, New Jersey
  - Research Site, Somerset, New Jersey
  - Research Site, Albany, New York
  - Research Site, Brooklyn, New York
  - Research Site, Clifton Park, New York
  - Research Site, Manhasset, New York
  - Research Site, New Windsor, New York
  - Research Site, New York, New York
  - Research Site, Staten Island, New York
  - Research Site, Stony Brook, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Charlotte, North Carolina
  - Research Site, Durham, North Carolina
  - Research Site, Greensboro, North Carolina
  - Research Site, Pinehurst, North Carolina
  - Research Site, Statesville, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Springfield, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Abington, Pennsylvania
  - Research Site, Camp Hill, Pennsylvania
  - Research Site, Hershey, Pennsylvania
  - Research Site, Horsham, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Charleston, South Carolina
  - Research Site, Ladson, South Carolina
  - Research Site, Lancaster, South Carolina
  - Research Site, Rapid City, South Dakota
  - Research Site, Jackson, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Tullahoma, Tennessee
  - Research Site, Allen, Texas
  - Research Site, Amarillo, Texas
  - Research Site, Cypress, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Katy, Texas
  - Research Site, Mansfield, Texas
  - Research Site, McKinney, Texas
  - Research Site, Odessa, Texas
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sherman, Texas
  - Research Site, Temple, Texas
  - Research Site, Tyler, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Falls Church, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Puyallup, Washington
  - Research Site, Seattle, Washington
  - Research Site, Tacoma, Washington
- Argentina (12):
  - Research Site, Buenos Aires
  - Research Site, CABA
  - Research Site, Ciudad de Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Esperanza
  - Research Site, Ganadero Baigorria
  - Research Site, Mar del Plata
  - Research Site, Rosario
  - Research Site, San Juan Bautista
  - Research Site, San Miguel de Tucumán
  - Research Site, Santa Fe
- Australia (10):
  - Research Site, Blacktown
  - Research Site, Cairns
  - Research Site, Canberra
  - Research Site, Chermside
  - Research Site, Clayton
  - Research Site, Concord
  - Research Site, Frankston
  - Research Site, Geelong
  - Research Site, Murdoch
  - Research Site, North Tamworth
- Austria (7):
  - Research Site, Braunau am Inn
  - Research Site, Graz
  - Research Site, Linz
  - Research Site, Saint Stefan/Stainz
  - Research Site, Salzburg
  - Research Site, Sankt Pölten
  - Research Site, Vienna
- Brazil (13):
  - Research Site, Aracaju
  - Research Site, Blumenau
  - Research Site, Brasília
  - Research Site, Campina Grande do Sul
  - Research Site, Campinas
  - Research Site, Curitiba
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, Rio de Janeiro
  - Research Site, São José dos Campos
  - Research Site, São Paulo
  - Research Site, Teresina
  - Research Site, Uberlândia
- Bulgaria (9):
  - Research Site, Botevgrad
  - Research Site, Dupnitsa
  - Research Site, Haskovo
  - Research Site, Kozloduy
  - Research Site, Pleven
  - Research Site, Plovdiv
  - Research Site, Sliven
  - Research Site, Sofia
  - Research Site, Stara Zagora
- Canada (23):
  - Research Site, New Westminster, British Columbia
  - Research Site, North Vancouver, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Sydney, Nova Scotia
  - Research Site, Cambridge, Ontario
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Newmarket, Ontario
  - Research Site, North York, Ontario
  - Research Site, Oakville, Ontario
  - Research Site, Oshawa, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Thunder Bay, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Chicoutimi, Quebec
  - Research Site, Greenfield Park, Quebec
  - Research Site, Montreal, Quebec
  - Research Site, Saint-Charles-Borromée, Quebec
  - Research Site, Saint-Jean-sur-Richelieu, Quebec
  - Research Site, Trois-Rivières, Quebec
- Chile (9):
  - Research Site, Antofagasta
  - Research Site, Punta Arenas
  - Research Site, Region Metropolitana
  - Research Site, San Bernardo
  - Research Site, Santiago
  - Research Site, Talcahuano
  - Research Site, Temuco
  - Research Site, Valdivia
  - Research Site, Victoria
- China (36):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chifeng
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hengyang
  - Research Site, Heze
  - Research Site, Hohhot
  - Research Site, Jinan
  - Research Site, Jining
  - Research Site, Lanzhou
  - Research Site, Liaocheng
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanchong
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Pingxiang
  - Research Site, Quzhou
  - Research Site, Sanya
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Ürümqi
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Xianyang
  - Research Site, Xuzhou
  - Research Site, Yangzhou
  - Research Site, Zhangjiakou
  - Research Site, Zunyi
- Colombia (8):
  - Research Site, Armenia
  - Research Site, Barranquilla
  - Research Site, Bogotá
  - Research Site, Cali
  - Research Site, Manizales
  - Research Site, Medellín
  - Research Site, Piedecuesta
  - Research Site, Rionegro
- Czechia (15):
  - Research Site, Brno
  - Research Site, Broumov
  - Research Site, Česká Lípa
  - Research Site, Jaroměř
  - Research Site, Louny
  - Research Site, Ostrava
  - Research Site, Pilsen
  - Research Site, Plzen - Bory
  - Research Site, Prague
  - Research Site, Přerov
  - Research Site, Slaný
  - Research Site, Svitavy
  - Research Site, Ustí Nad Labem
  - Research Site, Ústí nad Labem
  - Research Site, Zlín
- Finland (3):
  - Research Site, Helsinki
  - Research Site, Tampere
  - Research Site, Turku
- France (26):
  - Research Site, Béziers
  - Research Site, Bron
  - Research Site, Caen
  - Research Site, Cholet
  - Research Site, Créteil
  - Research Site, Dijon
  - Research Site, La Roche-sur-Yon
  - Research Site, La Tronche
  - Research Site, Le Coudray
  - Research Site, Limoges
  - Research Site, Meaux
  - Research Site, Montauban
  - Research Site, Montpellier
  - Research Site, Nantes
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Poitiers
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Rouen
  - Research Site, Saint-Quentin
  - Research Site, Strasbourg
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tours
  - Research Site, Valenciennes
- Germany (29):
  - Research Site, Bad Nauheim
  - Research Site, Bechhofen
  - Research Site, Berlin
  - Research Site, Bernau bei Berlin
  - Research Site, Chemnitz
  - Research Site, Coburg
  - Research Site, Dresden
  - Research Site, Elsterwerda
  - Research Site, Frankfurt
  - Research Site, Freiburg im Breisgau
  - Research Site, Goslar
  - Research Site, Göttingen
  - Research Site, Hagen
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Kaiserslautern
  - Research Site, Langen
  - Research Site, Leipzig
  - Research Site, Leverkusen
  - Research Site, Mainz
  - Research Site, Mönchengladbach
  - Research Site, Münster
  - Research Site, Paderborn
  - Research Site, Papenburg
  - Research Site, Regensburg
  - Research Site, Rostock
  - Research Site, Völklingen
  - Research Site, Wermsdorf
  - Research Site, Witten
- Greece (4):
  - Research Site, Athens
  - Research Site, Dragana
  - Research Site, Heraklio
  - Research Site, Thessaloniki
- Hungary (9):
  - Research Site, Balatonfüred
  - Research Site, Békéscsaba
  - Research Site, Budapest
  - Research Site, Gyula
  - Research Site, Hódmezővásárhely
  - Research Site, Kecskemét
  - Research Site, Orosháza
  - Research Site, Pécs
  - Research Site, Székesfehérvár
- India (19):
  - Research Site, Ahmedabad
  - Research Site, Ajmer
  - Research Site, Bangalore
  - Research Site, Belagavi
  - Research Site, Coimbatore
  - Research Site, Dehradun
  - Research Site, Delhi
  - Research Site, Hyderabad
  - Research Site, Kanpur
  - Research Site, Karamsad
  - Research Site, Kolkata
  - Research Site, Manipal
  - Research Site, Meerut
  - Research Site, Mysuru
  - Research Site, Nagpur
  - Research Site, New Delhi
  - Research Site, Pune
  - Research Site, Rudrapur
  - Research Site, Vijayawada
- Israel (12):
  - Research Site, Afula
  - Research Site, Ashkelon
  - Research Site, Beersheba
  - Research Site, Be’er Ya‘aqov
  - Research Site, Haifa
  - Research Site, Holon
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Nahariya
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tiberias
- Italy (13):
  - Research Site, Acquaviva delle Fonti
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Brescia
  - Research Site, Catania
  - Research Site, Catanzaro
  - Research Site, Cona
  - Research Site, Cortona
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Novara
  - Research Site, Pavia
  - Research Site, San Giovanni Rotondo
- Japan (43):
  - Research Site, Beppu-shi
  - Research Site, Bunkyō City
  - Research Site, Fujisawa-shi
  - Research Site, Fukui-shi
  - Research Site, Fukuoka
  - Research Site, Fukutsu-shi
  - Research Site, Hakusan-shi
  - Research Site, Higashiibaraki-gun
  - Research Site, Himeji
  - Research Site, Iwakuni-shi
  - Research Site, Kanazawa
  - Research Site, Kanonji-shi
  - Research Site, Kasuga-shi
  - Research Site, Kasugai-shi
  - Research Site, Kawaguchi
  - Research Site, Kawanishi-shi
  - Research Site, Kishiwada-shi
  - Research Site, Kitakyusyu-shi
  - Research Site, Kobe
  - Research Site, Kochi
  - Research Site, Kure-shi
  - Research Site, Maebashi
  - Research Site, Matsumoto-shi
  - Research Site, Meguro-ku
  - Research Site, Mito
  - Research Site, Moriyama-shi
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Ōita
  - Research Site, Sagamihara-shi
  - Research Site, Saitama Shi
  - Research Site, Saitama-shi
  - Research Site, Sakaishi
  - Research Site, Sakata
  - Research Site, Sanyoonoda-shi
  - Research Site, Toshima-ku
  - Research Site, Toyota
  - Research Site, Tsuchiura-shi
  - Research Site, Ueda-shi
  - Research Site, Uji-shi
  - Research Site, Uwajima-shi
  - Research Site, Yanagawa-shi
  - Research Site, Yokohama
- Malaysia (7):
  - Research Site, Kajang
  - Research Site, Kota Kinabalu
  - Research Site, Kota Samarahan
  - Research Site, Kuala Lumpur
  - Research Site, Kuala Terengganu
  - Research Site, Kuantan
  - Research Site, Sungai Buloh
- Mexico (17):
  - Research Site, Aguascalientes
  - Research Site, Chihuahua City
  - Research Site, Cuauhtémoc
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Mazatlán
  - Research Site, Metepec
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
  - Research Site, Morelia
  - Research Site, Querétaro
  - Research Site, San Luis Potosí City
  - Research Site, Tijuana
  - Research Site, Torreón
  - Research Site, Veracruz
  - Research Site, Xalapa
- Netherlands (6):
  - Research Site, Amsterdam
  - Research Site, Arnhem
  - Research Site, Emmen
  - Research Site, Goes
  - Research Site, Hardenberg
  - Research Site, Leeuwarden
- Peru (3):
  - Research Site, Bellavista
  - Research Site, Lima
  - Research Site, Piura
- Philippines (15):
  - Research Site, Angeles City
  - Research Site, Cebu City
  - Research Site, City of Taguig
  - Research Site, Davao City
  - Research Site, Iloilo City
  - Research Site, Las Piñas
  - Research Site, Mabalacat
  - Research Site, Makati
  - Research Site, Manadaluyong City
  - Research Site, Manila
  - Research Site, Marikina City
  - Research Site, Pasig
  - Research Site, Quezon City
  - Research Site, Roxas City
  - Research Site, West San Juan City
- Poland (24):
  - Research Site, Biała Podlaska
  - Research Site, Bielsko-Biala
  - Research Site, Bydgoszcz
  - Research Site, Chrzanów
  - Research Site, Gdansk
  - Research Site, Gdynia
  - Research Site, Katowice
  - Research Site, Kazimierza Wielka
  - Research Site, Kędzierzyn-Koźle
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Olsztyn
  - Research Site, Ostrów Mazowiecka
  - Research Site, Piekary Śląskie
  - Research Site, Poznan
  - Research Site, Rzeszów
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Tychy
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
- Romania (10):
  - Research Site, Afumaţi
  - Research Site, Arad
  - Research Site, Baia Mare
  - Research Site, Brasov
  - Research Site, Bucharest
  - Research Site, Cluj-Napoca
  - Research Site, Iași
  - Research Site, Satu Mare
  - Research Site, Târgu Mureş
  - Research Site, Timișoara
- Saudi Arabia (3):
  - Research Site, Dammam
  - Research Site, Jeddah
  - Research Site, Riyadh
- Slovakia (12):
  - Research Site, Banská Bystrica
  - Research Site, Bratislava
  - Research Site, Brezno
  - Research Site, Košice
  - Research Site, Martin
  - Research Site, Myjava
  - Research Site, Nitra
  - Research Site, Nové Zámky
  - Research Site, Považská Bystrica
  - Research Site, Prešov
  - Research Site, Rimavská Sobota
  - Research Site, Svidník
- South Africa (11):
  - Research Site, Bloemfontein
  - Research Site, Centurion
  - Research Site, Durban
  - Research Site, Johannesburg
  - Research Site, KwaDukuza
  - Research Site, Panorama
  - Research Site, Parow
  - Research Site, Pietermaritzburg
  - Research Site, Somerset West
  - Research Site, Soweto
  - Research Site, Worcester
- South Korea (15):
  - Research Site, Anyang-si
  - Research Site, Bucheon-si
  - Research Site, Busan
  - Research Site, Cheongju-si
  - Research Site, Daegu
  - Research Site, Daejeon
  - Research Site, Gwangju
  - Research Site, Gwangmyeong
  - Research Site, Incheon
  - Research Site, Junggu
  - Research Site, Seongnam-si
  - Research Site, Seoul
  - Research Site, Uijeongbu-si
  - Research Site, Wŏnju
  - Research Site, Yangsan
- Spain (7):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Lugo
  - Research Site, Madrid
  - Research Site, Majadahonda
  - Research Site, Seville
  - Research Site, Valencia
- Sweden (8):
  - Research Site, Alingsås
  - Research Site, Gothenburg
  - Research Site, Jönköping
  - Research Site, Karlstad
  - Research Site, Mölndal
  - Research Site, Stockholm
  - Research Site, Uppsala
  - Research Site, Västerås
- Taiwan (8):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yilan
  - Research Site, Yung Kang City
- Thailand (6):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Naimuang
  - Research Site, Pathum Thani
- Turkey (Türkiye) (13):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Dinar
  - Research Site, Eskişehir
  - Research Site, Istanbul
  - Research Site, Izmir
  - Research Site, Kocaeli
  - Research Site, Kütahya
  - Research Site, Merkez
  - Research Site, Muğla
  - Research Site, Sivas
- Ukraine (7):
  - Research Site, Chernivtsі
  - Research Site, Ivano-Frankivsk
  - Research Site, Kyiv
  - Research Site, Ternopil
  - Research Site, Uzhhorod
  - Research Site, Vinnytsia
  - Research Site, Zhytomyr
- United Kingdom (17):
  - Research Site, Airdrie
  - Research Site, Barnet
  - Research Site, Cambridge
  - Research Site, Clydebank
  - Research Site, Exeter
  - Research Site, Harefield
  - Research Site, Hastings
  - Research Site, High Wycombe
  - Research Site, Kent
  - Research Site, Kings Lynn
  - Research Site, Lincoln
  - Research Site, London
  - Research Site, Middlesbrough
  - Research Site, Portsmouth
  - Research Site, Sheffield
  - Research Site, Sunderland
  - Research Site, Wakefield
- Vietnam (10):
  - Research Site, Can Tho
  - Research Site, Da Nang
  - Research Site, Haiphong
  - Research Site, Hanoi
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City
  - Research Site, Hochiminh City
  - Research Site, Hochiminh
  - Research Site, Hồ Chí Minh
  - Research Site, Huế

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  "Yes", indicates that AZ are accepting requests for IPD, but this does not mean all requests will be approved.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA/PhRMA Data-Sharing Principles. For details of our timelines, please refer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. A Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- [Derived] Bhattacharya CS, Ericsson H, Johansson S, Parkinson J, Boca SM, Yang Y, Heijer M, Housler G, Leonsson-Zachrisson M, Hartleib-Geschwindner J, Pizzato PE. The effect of severe renal impairment on the pharmacokinetics, safety and tolerability of balcinrenone. Br J Clin Pharmacol. 2025 Jul;91(7):1937-1946. doi: 10.1002/bcp.70017. Epub 2025 Feb 17. PMID 39962632